CLINICAL TRIAL: NCT04611594
Title: Impact of Fluid Restriction in Patients With Pulmonary Congestion After Discharge From an Acute Decompensated Heart Failure Hospitalization: a Randomized Clinical Trial.
Brief Title: Fluid Restriction in Patients With Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Luis Eduardo Paim Rohde, Post Graduated Program of Federal University Program, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HCPA 2019-0216
Record Dates: First submitted 2020-09-15; First posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Heart Failure, Systolic; Heart Failure; With Decompensation; Pulmonary Congestion
Keywords: Pulmonary ultrasound; Fluid restriction; Water restriction; Congestion
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluid restriction (Experimental): Prescription to ingest approximately 20 ml / kg of ideal weight.
  Interventions: Behavioral: Fluid restriction
- Control (No Intervention): Prescription to ingest approximately 30 ml / kg of ideal weight, considered a normal amount of daily water intake.

INTERVENTIONS:
Behavioral: Fluid restriction — Ingestion of approximately 20 ml / kg of ideal weight,
  Arms: Fluid restriction

SUMMARY:
There is a concept increasingly consolidated by clinical evidence that at each hospitalization due to HF decompensation there is a substantial loss of quality of life, which is associated with an initial period of great clinical vulnerability, with high rates of rehospitalization and an increased risk of death. The non-pharmacological measures that are widely practiced and recommended for HF patients, such as fluid restriction, specially at the first 30 days after hospital discharge, still lack clearer evidence of their therapeutic efficacy.

DETAILED DESCRIPTION:
The need for hospitalization is an important marker of poor prognosis in patients with heart failure. It is estimated that 25% of patients presenting with acute heart failure are readmitted within 30 days. The maintenance of signs and symptoms of congestion at hospital discharge are common causes of hospital readmission. Thus, the reduction of these signs is a goal to be reached during hospitalization so that the chances of readmission are reduced. However, there is evidence that approximately ¼ of the patients are released despite persisting signs of congestive symptoms. It seems plausible to speculate that patients with HF at higher risk of rehospitalization would be those with the greatest chance of benefiting from therapeutic strategies that seek to reduce the congestive state, such as fluid restriction. In this scenario of initial vulnerability after hospitalization for acutely decompensated HF, recent studies have demonstrated a correlation in the number of B lines in the pulmonary ultrasound of patients at the time of hospital discharge and the prediction of frequent clinical outcomes. It was observed that the presence of pattern B, defined as the presence of more than 3 B lines in at least 2 pulmonary fields bilaterally, was associated with a worse prognosis (mortality from all causes and hospitalization due to decompensation). The present study, therefore, will evaluate the effect of outpatient fluid restriction on levels of NT-proBNP in patients who remain with signs of congestion based on pulmonary ultrasound at the bedside during hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Hospital admission for primary diagnosis of acutely decompensated heart failure, regardless of etiology, according to the criteria of the American College of Cardiology;
* Diagnosis on echocardiography of heart failure with reduced ejection fraction (<40%);
* Presence of pulmonary congestion defined as at least 2 pulmonary fields with more than 3 B lines in each field on pulmonary ultrasound at the time of hospital discharge.

Exclusion Criteria:

* Pulmonary fibrosis or other severe disease that changes the image acquisition (significant pleural effusion, severe pulmonary emphysema, previous pneumectomy or lobectomy, primary or metastatic lung cancer, breast implants);
* Pregnancy;
* Dialysis renal failure patient;
* Factors that could hinder follow-up (not returning to the outpatient clinic of Hospital de Clínicas);
* Disability or refusing to understand and adhere to the protocol;
* Refusal to sign consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
N-terminal pro-BNP | 30 days
  Variation in plasma NT pro-BNP levels (from the day of hospital discharge to approximately 30 days after).

SECONDARY OUTCOMES:
Pulmonary ultrasound | 30 days
  Variation in the total number of B lines in all lung fields measured by ultrasound (from the day of hospital discharge until approximately 30 days after).
Body weight | 30 days
  Variation of the patient's weight in kilograms (from the day of hospital discharge until approximately 30 days after)
Major cardiovascular and non-cardiovascular clinical events | 30 days
  Hospital admissions and death
Multidisciplinary clinical events related to heart failure | 30 days
  Six minutes walk test

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided